CLINICAL TRIAL: NCT03364504
Title: Biological Collection of Renal Cells for the Functional Study of the ABCC6 Transporter on iPS-derived Hepatocytes and Renal Cells
Brief Title: Biological Collection of Kidney Cells
Acronym: CRHiPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Université de Nantes (Other); Hungarian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 49RC17_0063
Record Dates: First submitted 2017-07-11; First posted 2017-12-06 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-06

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: PXE; renal cells; urine; calcification; omics; drug screening
MeSH Terms: conditions — Pseudoxanthoma Elasticum; Calcinosis | interventions — Urine Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PXE patients (Experimental): urine collection and culture of renal cells
  Interventions: Other: urine collection

INTERVENTIONS:
Other: urine collection — 3 urine collections during 24 hours

SUMMARY:
Our objective is to obtain human induced pluripotent stem cells from urine samples of PXE patients for further proteomic and metabolomic studies and treatment screening.

DETAILED DESCRIPTION:
Pseudoxanthoma elasticum (PXE) is a genetic multysystem disorder with cutaneous, ophtalmological and cardiovascular involvement.

PXE is associated with mutations of ABCC6 gene coding for the membrane transporter ABCC6 protein. This transporter is normally expressed in hepatocytes and epithelial cells of renal proximal convoluted tubules.

Thus, PXE could be regarded as a metabolic disease of hepatic and renal origin, with clinical and biological involvement/consequences for remote organs.

The substance transported by ABCC6 protein being still unknown, ethiological PXE treatment does not exist yet. However, ABCC6 deficiency is associated with low level of blood PPi (pyrophosphate), which is natural inhibitor of calcium-phosphate deposition.

The aim of the project is to obtain the renal cells derived from PXE patients for their further usage in proteomic and metabolomic studies, as well as for screening of treatment modalities aimed to correct ABCC6 functional deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patient with PXE diagnosed on clinical and histological criteria, according to current guidelines
* Patient aged over 18
* Patient informed, having understood the purpose and means of the study and signed the consent of participation
* Patient affiliated to the French social welfare system

Exclusion Criteria:

* Pregnant or nursing PXE woman
* Patient under guardianship, deprived of liberty by court or administrative decision, hospitalized without consent or admitted to a health or social institution for purposes other than research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Urine collection | 24 hours
  Three urine samples in each PXE in-patient consequences of the functional deficiency of the ABCC6 transporter involved in the pathophysiology of PXE

SECONDARY OUTCOMES:
Isolation and culture of renal cells | 8 weeks
  According to the routine procedure of our lab
Impact of ABCC6 mutations on renal cell functions | 3 months
  Proteomic and metabolomic and RNAseq approaches
High throughput screening of drugs to restore ABCC6 function in PXE patients renal cells | 3 months
  Evaluation of PPi release and other relevant readouts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Si-Tayeb K, Idriss S, Champon B, Caillaud A, Pichelin M, Arnaud L, Lemarchand P, Le May C, Zibara K, Cariou B. Urine-sample-derived human induced pluripotent stem cells as a model to study PCSK9-mediated autosomal dominant hypercholesterolemia. Dis Model Mech. 2016 Jan;9(1):81-90. doi: 10.1242/dmm.022277. Epub 2015 Nov 19. PMID 26586530
- [Result] Chassaing N, Martin L, Calvas P, Le Bert M, Hovnanian A. Pseudoxanthoma elasticum: a clinical, pathophysiological and genetic update including 11 novel ABCC6 mutations. J Med Genet. 2005 Dec;42(12):881-92. doi: 10.1136/jmg.2004.030171. Epub 2005 May 13. PMID 15894595
- [Result] Jansen RS, Duijst S, Mahakena S, Sommer D, Szeri F, Varadi A, Plomp A, Bergen AA, Oude Elferink RP, Borst P, van de Wetering K. ABCC6-mediated ATP secretion by the liver is the main source of the mineralization inhibitor inorganic pyrophosphate in the systemic circulation-brief report. Arterioscler Thromb Vasc Biol. 2014 Sep;34(9):1985-9. doi: 10.1161/ATVBAHA.114.304017. Epub 2014 Jun 26. PMID 24969777
- [Result] Jansen RS, Kucukosmanoglu A, de Haas M, Sapthu S, Otero JA, Hegman IE, Bergen AA, Gorgels TG, Borst P, van de Wetering K. ABCC6 prevents ectopic mineralization seen in pseudoxanthoma elasticum by inducing cellular nucleotide release. Proc Natl Acad Sci U S A. 2013 Dec 10;110(50):20206-11. doi: 10.1073/pnas.1319582110. Epub 2013 Nov 25. PMID 24277820